CLINICAL TRIAL: NCT05622409
Title: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Diffuse Glioma
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T3322
Record Dates: First submitted 2022-11-13; First posted 2022-11-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Primary Malignant Brain Tumors
Keywords: adult-type diffuse gliomas; next-generation sequencing; precision medicine
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. One H&E staining slide, and 15-20 tissue slides (5 um thickness) for cancer panel.
  2. Details of Tests/Collaborative Test Unit:
     Testing will take place in a certified precision medicine laboratory.
  3. Non-tumor Sample (Blood): Fifteen (15) ml of blood will be collected from the participant: 7 ml in EDTA tube (purple top) and 8 ml in Cell-Free DNA blood collection tube.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: Newly diagnosis arm (N=150): The study aims to obtain clinical information to correlate with genetic characterization of ATDGs of all types. Only patients with primary tumors that have recently received surgery are applicable.
- Arm 2: Post treatment arm 1 for training set (IDH-wild type ATDGs, N=50; IDH-mutant ATDGs, N=50): The study aims to compare the genetic differences of ATDGs in terms of IDH mutation status. Samples of primary tumors are preferred but can be replaced with recurrent ones. Paired samples are both eligible for typing if the recurrent diseases of IDH-mutant tumors possess potential altered genes (such as up grading per histology features).
- Arm 3: Post treatment arm 2 (recurrent ATDGs; N=25): The study will focus on recurrent diseases of ATDGs to study the consistency of genetic difference of the primary and the recurrent tumors. Tumor free is mandatory and needs to be documented after resection of the primary tumor. Patients remain eligible if IDH statuses are uncertain.

SUMMARY:
Glioma is a major histological subtype of primary malignant brain tumors in Taiwan, with distinct epidemiological, clinical, and pathological features comparing to the other common cancer diseases. The disease rarely appears with metastatic disease at diagnosis, and with the most malignant subtype, glioblastoma, occurs with preference in mid- to old-age. For decades, primary malignant brain tumors has been known as one of the most desperate disease without successful improvement regarding of the treatment. Surgical resection is the principle for the primary treatment of gliomas. Chemotherapy and radiotherapy are often applied to patients for adjuvant therapy of surgery to pursue the treatment effect. Disappointedly, vast majority of the patients would eventually develop disease recurrence, leaving only limited choice for salvage treatment thereafter. The prognosis of these patients remains desperate, and thus a better understanding of this deadly disease is crucial for finding better therapeutic strategies for these patients.

DETAILED DESCRIPTION:
With demand of molecular characterization in precise diagnosis, we proposed this registry study to explore the impact of the new criteria by applying next-generation sequencing. The specific aims of this project are (1) to establish the tumor genetic and molecular profiles of adult-type diffuse gliomas in Taiwan, (2) to understand the treatment prognosis depending on difference of the genetic and molecular profiles for adult-type diffuse gliomas in Taiwan, and (3) to reveal the evolutionary changes of genetic and molecular features of adult-type diffuse gliomas. The long-term goals of this study are to help implement personalized therapy, to develop novel therapy, and to improve outcomes of patients with adult-type diffuse gliomas. It is also expected to create a platform for data storage and sharing.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmation or suggestion of adult-type diffuse gliomas A. Diagnosis includes glioblastoma, astrocytoma, oligodendrocytoma that is listed in ATDG category per WHO criteria.

   B. Gliomas that are preferred as ATDGs from pathological and clinical views, but not given for confirmed diagnosis.
2. Willingness to provide archival or newly obtained tumor tissues for current study proposal.
3. Age equal or more than 20 years old (inform consent).
4. Life expectancy more than 3 months.
5. Patients fully understand the protocol with the willingness to have regular follow-up.
6. Additional criteria for individual arms A. [Arm 1] Within 2 months after surgery for primary tumor. B. [Arm 2] Total resection of primary tumors with tissue samples available for test.

C. [Arm 3] (1) Total resection of primary tumors with the paired primary and recurrent tissue samples available for test. (2) IDH test suggesting wild-type.

Exclusion Criteria:

1. Gliomas diagnosed or preferred as other categories than ATDGs, such as pediatric-type diffuse gliomas, circumscribed astrocytic gliomas, and others.
2. Inability to cooperate by providing a complete medical history.
3. Patients disagree to provide archived tumor samples.
4. Undesirable compliance.
5. Having a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Arm 1: (Newly diagnosis arm): Anticipated 100 patients. Arm 2: IDH expression (N=83 for IDH-mutant and N=82 for IDH-wild type) Arm 3:Recurrent and paired samples (N=10).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the genetic profiles in brain tumor patients in Taiwan. | 5 years
  ACTonco+ACTFusion Biospecimen Retention: Samples With DNA One H&E staining slide, and 15-20 tissue slides (5 um thickness) for cancer panel.
  Details of Tests/Collaborative Test Unit:
  Testing will take place in a certified precision medicine laboratory.
  Non-tumor Sample (Blood): Seven(7)ml of cell free DNA and Eight (8) ml of blood in EDTA tube will be collected from the participant

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Yu Chang, MD,PhD, Study Chair — National Health Research Institutes, Taiwan; Tsang-Wu Liu, MD, Study Chair — National Health Research Institutes, Taiwan; Yong-Kwang Tu, MD, PhD, Principal Investigator — Taipei Neuroscience Institute,Taipei Medical University
Locations (8):
- Taiwan (8):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University -Ministry of Health and Welfare Shuang-Ho Hospital, Taipei
  - CHANG GUNG MEMORIAL HOSPITAL, Linkou, Taoyuan District